CLINICAL TRIAL: NCT00762957
Title: A Multicenter, Double-Blind, Randomized, Placebo-Controlled, Parallel Study of the Safety and Efficacy of a Combination of TAK-559 and Metformin Compared to Placebo and Metformin in the Treatment of Patients With Type 2 Diabetes Mellitus
Brief Title: Safety and Efficacy of TAK-559 in Combination With Metformin in Patients With Type 2 Diabetes Mellitus.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Hepatic Safety Signal Identified.
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 01-04-TL-559-029; U1111-1128-4945 (Registry Identifier: WHO)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2012-02-28 (Estimated); Status verified 2012-02

CONDITIONS: Diabetes Mellitus
Keywords: Glucose Metabolism Disorder; Dysmetabolic Syndrome; Type II Diabetes; Diabetes Mellitus, Lipoatrophic; Dyslipidemia; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus; Glucose Metabolism Disorders; Diabetes Mellitus, Type 2; Diabetes Mellitus, Lipoatrophic; Dyslipidemias | interventions — (E)-4-(4-((5-methyl-2-phenyl-1,3-oxazol-4-yl)methoxy)benzyloxyimino)-4-phenylbutyric acid; Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- TAK-559 16 mg QD + Metformin QD (Experimental)
  Interventions: Drug: TAK-559 and metformin
- TAK-559 32 mg QD + Metformin QD (Experimental)
  Interventions: Drug: TAK-559 and metformin
- Metformin QD (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: TAK-559 and metformin — TAK-559 16 mg, tablets, orally, once daily and metformin stable dose orally, once daily for up to 26 weeks.
  Arms: TAK-559 16 mg QD + Metformin QD
Drug: TAK-559 and metformin — TAK-559 32 mg, tablets, orally, once daily and metformin stable dose, orally, once daily for up to 26 weeks.
  Arms: TAK-559 32 mg QD + Metformin QD
Drug: Metformin — TAK-559 placebo-matching tablets, orally, once daily and metformin stable dose, orally, once daily for up to 26 weeks.
  Arms: Metformin QD

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of TAK-559, once daily (QD), taken in combination with metformin in treating subjects with type 2 diabetes mellitus

DETAILED DESCRIPTION:
Insulin is a primary regulator of blood glucose concentrations. A subnormal response to circulating insulin levels at target tissues leads to a decrease in insulin-mediated glucose uptake. Insulin resistance is associated with normal to high insulin levels and is often accompanied by dyslipidemia, a disruption in lipid metabolism resulting in increased triglycerides and low-density lipoprotein levels as well as decreased high-density lipoprotein levels in patients with type 2 diabetes mellitus. In the early stages of insulin resistance, a compensatory mechanism of increased insulin secretion by the pancreas maintains normal to near-normal glucose levels. Once the pancreas fails to maintain the increased insulin output, overt type 2 diabetes mellitus occurs.

Insulin also plays an important role in the metabolism of fat and proteins and exerts its influence at the peroxisome proliferator-activated receptor level. Peroxisome proliferator-activated receptor -alpha receptors are expressed predominantly in skeletal muscle, adipose tissue, heart, liver, kidney, gut, macrophages, and vascular tissue, and play a key role in energy storage, glucose homeostasis, and vascular biology. Thus, as insulin activates peroxisome proliferator-activated receptor-alpha receptors, this results in the cellular uptake of glucose. Peroxisome proliferator-activated receptor receptors are ligand-activated transcription elements that regulate gene expression necessary for metabolism. For this reason, peroxisome proliferator-activated receptors play a pivotal role in glucose homeostasis, adipocyte differentiation, and lipid storage. The genes predominantly targeted by transcription activity of activated peroxisome proliferator-activated receptor-alpha receptors are those that mediate fatty acid uptake, fatty acid oxidation, and lipoprotein metabolism. As such, peroxisome proliferator-activated receptor-alpha agonists have their greatest effect on lipid metabolism and vascular biology.

TAK-559 is a novel oxyiminoalkanoic acid under investigation for use as an oral agent in the treatment of patients with type 2 diabetes mellitus. TAK-559 has partial peroxisome proliferator-activated receptor-alpha agonist activity, potent peroxisome proliferator-activated receptor-alpha activity, and modest peroxisome proliferator-activated receptor-gamma activity at high concentrations in nonclinical models.

This study was designed to evaluate the safety and glycemic control of TAK-559 in patients with type 2 diabetes mellitus taking metformin for whom monotherapy with an oral anti-diabetic had been insufficient.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 2 diabetes mellitus, and on a stable dose of an oral antidiabetic monotherapy before Screening A.
* Female patients of childbearing potential who were sexually active agreed to use adequate contraception, and could neither pregnant nor lactating from Screening throughout the duration of the study.
* Had a glycosylated hemoglobin level greater than or equal to 8.0% and less than or equal to 10.0% at Screening B.
* Had a fasting plasma glucose greater than or equal to 126 mg/dL (7.0 mmol/L) at Screening B.
* Taking a stable dose of at least 1000 mg of metformin for at least 30 days before Screening B.
* Had a stable or worsening self-monitoring blood glucose level while taking metformin.
* Had a low-density lipoprotein less than 160 mg/dL (4.1 mmol/L) at Screening A.
* Had a body mass index was less than or equal to 45 kg/m2 at Screening A.
* Was willing to be counseled by the investigator or designee to follow an individualized, weight-maintaining diet during the study period.
* Had evidence of insulin secretory capacity as demonstrated by a C-peptide concentration of greater than or equal to 1.5 ng/mL (0.50 nmol/L) at Screening A, and if necessary, after a repeat at Screening B.
* Was able to perform daily self-monitoring blood glucose tests throughout the study.
* Had a normal thyroid-stimulating hormone level of less than 5.5 μIU/mL (5.5 mIU/L) and greater than or equal to 0.35 μIU/mL (0.35 mIU/L) at Screening A.
* Was in good health as determined by a physician (ie, via medical history and physical examination), other than a diagnosis of type 2 diabetes mellitus.
* Had fasting clinical laboratory results within the normal ranges for the testing laboratory, or if not, the results were deemed not clinically significant by the investigator before Randomization.

Exclusion Criteria:

* Diagnosed with type 1 diabetes mellitus, hemochromatosis, or had a history of ketoacidosis.
* Had any condition known to invalidate glycosylated hemoglobin results (eg, hemolytic states or hemoglobinopathies).
* Took any disallowed medication, prescription medication, herbal treatment or over-the counter medication that may have interfered with evaluation of the study medication, including:

  * Insulin
  * Oral antidiabetics including sulfonylureas and alpha-glucosidase inhibitors
  * Systemic corticosteroids
  * Warfarin
  * Rifampin
  * St. John's Wort.
  * Thiazolidinediones
  * Peroxisome proliferator-activated receptor agonists
  * Nicotinic Acid
  * Fibrates
* Had a history of myocardial infarction, coronary angioplasty or bypass graft, unstable angina pectoris, transient ischemic attacks, clinically significant abnormal electrocardiogram, or documented cerebrovascular accident within 6 months before Screening A.
* Had abdominal, thoracic, or vascular surgery within 6 months before Screening A that in the investigator's opinion warranted exclusion from the study.
* Had a creatine phosphokinase value greater than 3 times the upper limit of normal at Screening A.
* Had persistent unexplained microscopic or macroscopic hematuria or a history of bladder cancer.
* Had a triglyceride level greater than 500 mg/dL (5.6 mmol/L) at Screening A.
* Received any alteration in allowed lipid lowering medication (dose or drug) within 2 months of Randomization, if applicable. The patient remained on a stable dose throughout the study. If deemed necessary, the dose could have been lowered with prior approval from the Sponsor.
* Donated and/or received any blood or blood products within 3 months before Randomization.
* Had a history of drug abuse or a history of alcohol abuse within 2 years before Randomization
* Had a systolic blood pressure greater than 140 mm Hg or a diastolic blood pressure of greater than 95 mm Hg at Screening B.
* Had significant cardiovascular disease including but not limited to, New York Heart Association Functional (Cardiac) Classification III or IV.
* Had a history of cancer other than basal cell or stage 1 squamous cell carcinoma of the skin that had not been in remission within 5 years before Randomization.
* Had an alanine aminotransferase or aspartate aminotransferase level greater than 3 times the upper limit of normal, active liver disease, or jaundice at Screening A.
* Had a positive anti-hepatitis B surface antigen, or anti-hepatitis B e antigen test results at Screening A.
* Was currently taking another investigational study medication or had taken an investigational study medication within 30 days before Screening A.
* Had any other serious disease or condition at Screening A or at Randomization that might have affected life expectancy or made it difficult to successfully manage and follow the patient according to the protocol.

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2004-11; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Final Visit.

SECONDARY OUTCOMES:
Change from baseline in glycosylated hemoglobin. | Weeks 2, 4, 8, 12, 16 and 20
Change from baseline in fasting plasma glucose. | Weeks 2, 4, 8, 12, 16, 20 and Final Visit
Change from baseline in serum insulin. | Weeks 4, 12, 16, 20 and Final Visit.
Change from baseline in C-peptide. | Weeks 4, 12, 16, 20 and Final Visit.
Change from baseline in triglycerides. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in total cholesterol. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in high-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in low-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in very-low-density lipoprotein. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in apolipoproteins A1 and B 100. | Final Visit
Change from baseline in free fatty acids. | Weeks 12, 16, 20 and Final Visit.
Change from baseline in thrombosis marker plasminogen activator inhibitor-1 | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in thrombosis marker fibrinogen. | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in inflammation marker Interleukin-6. | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in inflammation marker C-reactive protein. | Weeks 4, 12, 16, 20 and Final Visit
Change from baseline in urinary albumin to creatinine ratio. | Weeks 12, 16, 20 and Final Visit

CONTACTS AND LOCATIONS:
Overall Officials: VP Biological Sciences, Study Director — Takeda